CLINICAL TRIAL: NCT02357069
Title: Multi-center (in Korea and Japan), Double-blind, Randomized, Parallel-group Study to Evaluate Similarity of Efficacy and Safety of LBEC0101 50mg Subcutaneous Weekly Injection to Enbrel® 50mg Subcutaneous Weekly Injection, as Adjunctive Therapy to Methotrexate (MTX), in Patients With Active Rheumatoid Arthritis Who Had an Inadequate Response to MTX
Brief Title: A Study Comparing LBEC0101 to Enbrel® in Subjects With Active Rheumatoid Arthritis Despite Methotrexate Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LG Life Sciences (Industry)
Collaborators: Mochida Pharmaceutical Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-ECCL002
Record Dates: First submitted 2015-01-29; First posted 2015-02-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; LBEC0101

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- LBEC0101 (Experimental): Etanercept
  Interventions: Drug: LBEC0101
- Enbrel (Active Comparator): Etanercept
  Interventions: Drug: Enbrel

INTERVENTIONS:
Drug: Enbrel — Etanercept
  Arms: Enbrel
Drug: LBEC0101 — Etanercept
  Arms: LBEC0101

SUMMARY:
This is a randomized, double-blind, parallel group, multicenter clinical study to evaluate the efficacy, safety, pharmacokinetics and immunogenicity of LBEC0101 compared to Enbrel in subjects with active Rheumatoid Arthritis despite Methotrexate therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients from 20 years to 75 years of age when signing Informed Consent.
* Diagnosed as having RA according to the revised 1987 ACR criteria for at least 6 months prior to screening
* Patients who have inadequate response to MTX administered for at least 12 weeks before the beginning of screening period and on a stable dose.

Exclusion Criteria:

* patients with active tuberculosis or latent tuberculosis based on current clinical symptoms, chest X-ray test and IFN-γ release assay at screening
* patients with any of the following concomitant diseases and/or history within 24 weeks before the first administration of investigational products in this study; Serious infectious disease, Opportunistic infection, Chronic or recurrent infectious disease
* patients with any seropositive result for hepatitis B or hepatitis C or HIV
* patients who have any of the following diseases; Sepsis, Demyelinating disorders, Lymphoproliferative disease, Infection with prosthetic joint, Autoimmune diseases other than rheumatoid arthritis

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Disease activity score based on a 28 joint count (DAS28) | Week 24

CONTACTS AND LOCATIONS:
Locations (2):
- Mochida Investigational site, Tokyo, Japan
- LGLS Investigational site, Seoul, South Korea

REFERENCES:
- [Derived] Matsuno H, Tomomitsu M, Hagino A, Shin S, Lee J, Song YW. Phase III, multicentre, double-blind, randomised, parallel-group study to evaluate the similarities between LBEC0101 and etanercept reference product in terms of efficacy and safety in patients with active rheumatoid arthritis inadequately responding to methotrexate. Ann Rheum Dis. 2018 Apr;77(4):488-494. doi: 10.1136/annrheumdis-2017-212172. Epub 2017 Dec 19. PMID 29259050